CLINICAL TRIAL: NCT04006080
Title: Investigation of the Faecal Loss of Vedolizumab and Its Role in Influencing Serum Drug Levels, Outcomes and Response in Ulcerative Colitis
Acronym: FAVOUR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002794-21
Record Dates: First submitted 2019-02-13; First posted 2019-07-02 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vedolizumab (Experimental)
  Interventions: Biological: Vedolizumab

INTERVENTIONS:
Biological: Vedolizumab — Intravenously administered selective leukocyte adhesion molecule inhibitor
  Other Names: Entyvio

SUMMARY:
The purpose of this study is to study the loss of vedolizumab in stool in patients with active ulcerative colitis (UC).

Patients with moderate-to-severe UC who are commencing induction therapy with vedolizumab will be enrolled into a prospective study and stool will be collected for faecal vedolizumab measurement at days 1, 4 and 7; and again at weeks 2, 6 and 14. They will also be evaluated at three time-points (weeks 2, 6 and 14) for clinical and biochemical UC disease activity as well as serum vedolizumab concentrations and anti-vedolizumab antibodies.

DETAILED DESCRIPTION:
Primary objective

- To determine whether vedolizumab is present in significant quantities in the stool of patients receiving induction therapy with vedolizumab for active UC.

Secondary objective (s)

* To evaluate whether the presence and quantity of vedolizumab in stool can be used to predict primary non-response to vedolizumab.
* To explore whether a correlation exists between stool vedolizumab concentrations, serum vedolizumab concentrations and UC disease activity and extent.
* To determine whether there is a correlation between stool and serum vedolizumab levels and trafficking of Th1/Th17 effector memory CD4+ T-cells (the key pathogenic subset in IBD) to the colon in UC.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over, either male or female
* Moderate-to-severe UC, defined as:

  - SCCAI > 5 and, i. A raised fecal calprotectin (> 59 μg/g) or, ii. A raised CRP (> 5 mg/L) or, iii. Endoscopic disease activity Mayo 2 or above, Evaluated within 6 weeks of study enrollment
* Commencing vedolizumab treatment
* Sufficient English language skills to understand the patient information sheet and consent form

Exclusion Criteria:

* Contra-indication to vedolizumab (i.e. known serious or severe hypersensitivity reaction to vedolizumab or any of its excipients)
* Imminent need for colectomy (i.e. colectomy is being planned)
* Previous ileoanal pouch formation
* Active severe infections such as tuberculosis, sepsis, cytomegalovirus, listeriosis, and opportunistic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in vedolizumab concentrations in stool | Days 1, 4 and 7; and weeks 2, 6 and 14
  Evaluated using an enzyme-linked immunosorbent assay (ELISA)

SECONDARY OUTCOMES:
UC endoscopic activity | Baseline and week 14
  Evaluated using the Mayo Endoscopic Score: Mayo 0 = normal; Mayo 1= mild inflammation; Mayo 2 = moderate inflammation; Mayo 3 = severe inflammation
UC endoscopic activity | Baseline and week 14
  Evaluated using the Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score: Vascular pattern= Normal (0), patchy loss (1), obliterated (2); Bleeding = None (0), mucosal (1), luminal mild (2), luminal moderate (3); Erosions/ulcers = None (0), erosions (1), superfical ulcer (2), deep ulcer (3)
Clinical UC disease activity | Day 0, weeks 2, 6 and 14
  Evaluated using Patient Reported Outcome 2 (PRO2) Questionnaire: Stool frequency= normal (0), 1-2 more (1), 3-4 more (2), 5 or more stools than normal (3); Rectal bleeding= no blood (0), streaks of blood <50% time (1), obvious blood >50% time (2), blood alone passes (3)
Vedolizumab serum concentrations | Weeks 2, 6 and 14
  Evaluated using a drug-sensitive enzyme-linked immunosorbent assay (ELISA)
Vedolizumab anti-drug antibody levels | Weeks 2, 6 and 14
  Evaluated using a drug-sensitive enzyme-linked immunosorbent assay (ELISA)
Faecal calprotectin | Day 0, weeks 2, 6 and 14
  Evaluated using a drug-sensitive enzyme-linked immunosorbent assay (ELISA)
Serum CRP (mg/L) | Day 0, weeks 2, 6 and 14
Serum albumin (g/L) [40-52g/L] | Day 0, weeks 2, 6 and 14
Quality of life questionnaire | Day 0, weeks 2, 6 and 14
  IBD-Control questionnaire
Clinical UC disease activity | Day 0, weeks 2, 6 and 14
  Evaluated using the Simple Clinical Colitis Activity Index score: Bowel frequency day= 0-3 (0), 4-6 (1), 7-9 (2), >9 (3); Bowel frequency night= 0 (0), 1-3 (1), 4-6 (2); Urgency of defectation= None(0), Hurry (1), immediately (2), incontinence (3); Blood in stool = None (0), trace (1), occasional frank (2), usually frank (3); General well being= very well (0), slightly below par (1), poor (2), very poor (3), terrible (4); Extracolonic features (1 point for each) = arthritis, uveitis, erythema nodosum, pyoderma gangrenosum. Remission SCCAI ≤ 2; Response SCCAI ≤ 5, with a decrease by ≥ 2; Relapse SCCAI ≥ 5 (following a response)
UC histological activity | Day 0 and week 14
  Evaluated using Nancy Histological Index

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Haens G, Sandborn WJ, Feagan BG, Geboes K, Hanauer SB, Irvine EJ, Lemann M, Marteau P, Rutgeerts P, Scholmerich J, Sutherland LR. A review of activity indices and efficacy end points for clinical trials of medical therapy in adults with ulcerative colitis. Gastroenterology. 2007 Feb;132(2):763-86. doi: 10.1053/j.gastro.2006.12.038. Epub 2006 Dec 20. No abstract available. PMID 17258735
- [Background] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Background] Travis SP, Schnell D, Krzeski P, Abreu MT, Altman DG, Colombel JF, Feagan BG, Hanauer SB, Lichtenstein GR, Marteau PR, Reinisch W, Sands BE, Yacyshyn BR, Schnell P, Bernhardt CA, Mary JY, Sandborn WJ. Reliability and initial validation of the ulcerative colitis endoscopic index of severity. Gastroenterology. 2013 Nov;145(5):987-95. doi: 10.1053/j.gastro.2013.07.024. Epub 2013 Jul 25. PMID 23891974
- [Background] Jairath V, Khanna R, Zou GY, Stitt L, Mosli M, Vandervoort MK, D'Haens G, Sandborn WJ, Feagan BG, Levesque BG. Development of interim patient-reported outcome measures for the assessment of ulcerative colitis disease activity in clinical trials. Aliment Pharmacol Ther. 2015 Nov;42(10):1200-10. doi: 10.1111/apt.13408. Epub 2015 Sep 21. PMID 26388424
- [Background] Travis SP, Schnell D, Krzeski P, Abreu MT, Altman DG, Colombel JF, Feagan BG, Hanauer SB, Lemann M, Lichtenstein GR, Marteau PR, Reinisch W, Sands BE, Yacyshyn BR, Bernhardt CA, Mary JY, Sandborn WJ. Developing an instrument to assess the endoscopic severity of ulcerative colitis: the Ulcerative Colitis Endoscopic Index of Severity (UCEIS). Gut. 2012 Apr;61(4):535-42. doi: 10.1136/gutjnl-2011-300486. Epub 2011 Oct 13. PMID 21997563
- [Background] Bodger K, Ormerod C, Shackcloth D, Harrison M; IBD Control Collaborative. Development and validation of a rapid, generic measure of disease control from the patient's perspective: the IBD-control questionnaire. Gut. 2014 Jul;63(7):1092-102. doi: 10.1136/gutjnl-2013-305600. Epub 2013 Oct 9. PMID 24107590
- [Background] Marchal-Bressenot A, Salleron J, Boulagnon-Rombi C, Bastien C, Cahn V, Cadiot G, Diebold MD, Danese S, Reinisch W, Schreiber S, Travis S, Peyrin-Biroulet L. Development and validation of the Nancy histological index for UC. Gut. 2017 Jan;66(1):43-49. doi: 10.1136/gutjnl-2015-310187. Epub 2015 Oct 13. PMID 26464414
- [Background] Globig AM, Hennecke N, Martin B, Seidl M, Ruf G, Hasselblatt P, Thimme R, Bengsch B. Comprehensive intestinal T helper cell profiling reveals specific accumulation of IFN-gamma+IL-17+coproducing CD4+ T cells in active inflammatory bowel disease. Inflamm Bowel Dis. 2014 Dec;20(12):2321-9. doi: 10.1097/MIB.0000000000000210. PMID 25248005